CLINICAL TRIAL: NCT02018224
Title: Achilles Tendon Rupture, Comparison Two Different Operative Techniques. Prospective Randomized Controlled Trial. 14 Years Follow-up.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: evo-rad-akilles3
Record Dates: First submitted 2013-11-27; First posted 2013-12-23 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture, operative treatment, elongation, long-term follow up.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- End-to-end suturation without augmentation (Experimental)
  Interventions: Procedure: End-to-end suturation without augmentation
- End-to-end suturation with augmentation (Experimental)
  Interventions: Procedure: End-to-end suturation with augmentation.

INTERVENTIONS:
Procedure: End-to-end suturation without augmentation — End-to-end suturation without augmentation; Irregular tendon ends were cleaned and repaired by the Krackow technique with two separate 0-gauge absorbable sutures.
  Arms: End-to-end suturation without augmentation
Procedure: End-to-end suturation with augmentation. — End-to-end suturation with augmentation; End-to-end suturation as above with a 10 mm wide central gastrocnemius aponeurosis flap, as proposed by Silfverskjöld.
  Arms: End-to-end suturation with augmentation

SUMMARY:
The intention is to compare 60 patients with Achilles tendon rupture, who where randomized in 1998-2001 preoperatively to receive end-to-end suturation by the Krackow locking loop technique either without augmentation or with one central down-turned gastrocnemius fascia flap (Silfverskjöld). Postoperative care was identical for both groups; A brace allowed free active plantar flexion of the ankle postoperatively, whereas dorsiflexion was restricted to neutral for the first three weeks. Weight bearing was limited for six weeks. To compare these treatments, we use 1998 published Leppilahti-score, Rand-36 quality of life-questionnaire and MRI. Mean follow-up time is 14 years.

Hypothesis; Augmentation with a down-turned gastrocnemius fascia flap does not provide better result than would end-to-end suture repair with use of the Krackow locking loop surgical technique in long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Total achilles tendon rupture diagnose.

Exclusion Criteria:

* more than 7 days old rupture, local corticosteroids injection in around the achilles tendon, rupture was open/ there where skin problems over achilles tendon area, patient lived abroad, if the main author was unavailable, or patient refused to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 1998-10; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Subjective results in conservative and operative treatment of Achilles tendon rupture. | 14 years
  Subjective results consists of Rand-36 questionnaire and part of Leppilahti-scores questionnaire.
Objective results in operative treatment of Achilles tendon rupture. | 14 years
  Objective results consists of calf muscle isokinetic strength measurements and MRI-findings.

SECONDARY OUTCOMES:
Achilles tendon MRI-findings in operative and conservative treatment of achilles tendon rupture | 14 years
  We study calf muscle volume, achilles tendon volume, fat degeneration and achilles tendon elongation.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland